CLINICAL TRIAL: NCT06418386
Title: Clinical Assessment of Antimicrobial Effect of Rotary Versus Manual Filing System Using Different Irrigants in Primary Molars
Brief Title: Bacterial Reduction of Rotary Versus Manual Filing System Using Different Irrigants in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Menna Mahgoub, principle investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M18060722
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Necrotic Pulp
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Intervention Model Description: The children will be randomly divided into 2 main groups according to type of file used in root canal preparation:
  Group I with manual file. Group II with rotary file.
  Then the children will be randomly sub grouped according to irrigant that will be used:
  Group IA and group II A with normal saline. Group IB and group II B with neem . Group IC and group II C with NaOCl
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- manual saline (Active Comparator): manual k files for pulpectomy and normal saline irrigation
  Interventions: Procedure: manual saline IA
- manual neem extract (Experimental): manual k files and 100% neem extract
  Interventions: Procedure: manual neem IB
- manual sodium hypochlorite (Experimental): mannul k files and 1% sodium hypochlorite
  Interventions: Procedure: manual sodium hypochlorite IC
- rotary saline (Experimental): AF baby files for pediatric( fanta ) and normal saline
  Interventions: Procedure: rotary saline IIA
- rotary neem (Experimental): AF baby files for pediatric( fanta ) and 100% NEEM EXTRACT
  Interventions: Procedure: rotary neem IIB
- rotary sodium hypochloride (Experimental): AF baby files for pediatric( fanta ) and 1% sodium hypochloride
  Interventions: Procedure: rotary sodoium hypochlorite IIC

INTERVENTIONS:
Procedure: manual saline IA — * The procedural tooth is anesthetized and isolated with rubber dam. The tooth and adjacent rubber dam will be disinfected with tincture of iodine solution, All carious tissue will be removed by hight speed handpiece, distal cannel of mandibular primary molars and palatal cannel of maxillary primary molars will be chosen for sampling procedure.
  * A sterile broach will be inserted to obtain root cannel content then sterile paper point inserted to root canal and will be left for 1 min ,The paper point will be removed with sterilized tweezer which will immediately transferred to tube containing transport medium (eppendrof of containing 200 μl nutrient broth medium),using manual k file starting with #15 and irrigation with normal saline
  * Post irrigation sample and pre-preparation sample will be transferred to microbiological laboratory Canals will be filed with obturation material(Metapex)then crown will be restored with glass inomar and stainless steel crown
  Arms: manual saline
Procedure: manual neem IB — * The procedural tooth is anesthetized and isolated with rubber dam. The tooth and adjacent rubber dam will be disinfected with tincture of iodine solution
  * . All carious tissue will be removed by high speed hand piece
    , distal cannel of mandibular primary molars and palatal cannel of maxillary primary molars will be chosen for sampling procedure.
  * A sterile broach will be inserted to obtain root cannel content then sterile paper point inserted to root canal and will be left for 1 min 19 The paper point will be removed with sterilized tweezer which will immediately transferred to tube containing transport medium (eppendrof of containing 200 μl nutrient broth medium).
  * using manual file and irrigation with neem leaf extract 100%
  * Post irrigation sample and pre-preparation sample will be transferred to microbiological laboratory Canals will be filed with obturation material(Metapex)then crown will be restored with glass inomar and stainless steel crown
  Arms: manual neem extract
Procedure: manual sodium hypochlorite IC — * adjacent rubber dam will be disinfected with tincture of iodine solution
  * . All carious tissue will be removed by hight speed hand piece
  * distal cannel of mandibular primary molars and palatal cannel of maxillary primary molars will be chosen for sampling procedure.
  * A sterile broach will be inserted to obtain root cannel content then sterile paper point inserted to root canal and will be left for 1 min 19 The paper point will be removed with sterilized tweezer which will immediately transferred to tube containing transport medium (eppendrof of containing 200 μl nutrient broth medium).
  * using manual file and irrigation with 1% sodium hypochlorite
  * Post irrigation sample and pre-preparation sample will be transferred to microbiological laboratory Canals will be filed with obturation material(Metapex)then crown will be restored with glass inomar and stainless steel crown
  Arms: manual sodium hypochlorite
Procedure: rotary saline IIA — * shaping and cleaning done with using AF baby fanta files open file:#17 taper 08,then #20 taper 04 ,yellow then #25 taper 04 red , then #30 taper 04 blue . the files activated with torque 2 and speed 350 . Irrigation with normal saline
  * Post irrigation sample and pre-preparation sample will be transferred to microbiological laboratory Canals will be filed with obturation material(Metapex)then restored with glass inomar and stainless steel crown
  Arms: rotary saline
Procedure: rotary neem IIB — * The procedural tooth is anesthetized and isolated with rubber dam as mentioned
  * All carious tissue will be removed by high speed hand piece ,distal cannel of mandibular primary molars and palatal cannel of maxillary primary molars will be chosen for sampling procedure.
  * A sterile broach will be inserted to obtain root cannel content then sterile paper point inserted to root canal and will be left for 1 min The paper point will be removed with sterilized tweezer which will immediately transferred to tube containing transport medium (eppendrof of containing 200 μl nutrient broth medium).
  * using AF baby fanta files SAME AS METION BEFORE ,and irrigation with 100%neem extract
  * Post irrigation sample and pre-preparation sample will be transferred to microbiological laboratory Canals will be filed with obturation material(Metapex)then crown will be restored with glass inomar and stainless steel crown
  Arms: rotary neem
Procedure: rotary sodoium hypochlorite IIC — * The procedural tooth is anesthetized and isolated with rubber dam as mentioned
  * All carious tissue will be removed by hight speed hand piece,distal cannel of mandibular primary molars and palatal cannel of maxillary primary molars will be chosen for sampling procedure.
  * A sterile broach will be inserted to obtain root cannel content then sterile paper point inserted to root canal and will be left for 1 min The paper point will be removed with sterilized tweezer which will immediately transferred to tube containing transport medium (eppendrof of containing 200 μl nutrient broth medium).
  * using AF baby fanta files SAME AS MENTION BEFORE , and irrigation with 1% sodium hypochlorite
  * Post irrigation sample and pre-preparation sample will be transferred to microbiological laboratory Canals will be filed with obturation material(Metapex)then crown will be restored with glass inomar and stainless steel crown
  Arms: rotary sodium hypochloride

SUMMARY:
This study will evaluate and compare the microbial efficacy of rotary and manual filing system using Neem extract, NaOCL and saline . with hypotheses that neem can used alternative to sodium hypochlorite and there is no difference between rotary and manual filling in bacterial reduction.

DETAILED DESCRIPTION:
The calculated sample size of the study will be 22 participants for each group at 5% level of significance and 80 % power 30 participants for each group (10 for The sample size will be increased tocompensate for incomplete data and to increase the study each subgroup) topower

Grouping:

30 child will be selected from the Pediatric Clinic, Faculty of Dentistry, Mansoura University .the child should have 2 contralateral primary molars indicated for pulpectomy. The children will be randomly divided into 2 main groups according to type of file used in root canal preparation: Group I with manual file. Group II with rotary file.

Then the children will be randomly sub grouped according to irrigant that will be used:

Group IA and group II A with normal saline. Group IB and group II B with neem . Group IC and group II C with NaOCl . clinical procedures :

1. Psychological management of child
2. X-ray for inclusion criteria
3. The procedural tooth is anesthetized and isolated with rubber dam. The tooth and adjacent rubber dam will be disinfected with tincture of iodine solution
4. . All carious tissue will be removed by sterilized round bur and root canal access will be done
5. On gaining the access, distal cannel of mandibular primary molars and palatal cannel of maxillary primary molars will be chosen for sampling procedure.
6. A sterile broach will be inserted to obtain root cannel content then sterile paper point inserted to root canal and will be left for 1 min 19 The paper point will be removed with sterilized tweezer which will immediately transferred to tube containing transport medium (eppendrof of containing 200 μl nutrient broth medium).
7. In-group 1 will be prepared with manual files the irrigation with saline in IA, with neem in IB and irrigation with NaOCl in IC.
8. In group II will be prepared with rotary files the irrigation with saline in IIA, with neem in IIB, with NaOCl in IIC
9. The sterile paper point will be introduced into root cannel and will be left for 1 min, the paper point will be removed with sterilized tweezer and then transferred to a tube containing transport medium 19.
10. Post irrigation sample and pre-preparation sample will be transferred to microbiological laboratory.
11. Canals will be filed with obturation material(Metapex)then crown will be restored with glass inomar and stainless steel crown

Laboratory procedures :

1. All samples will be incubated on blood agar aerobically and anaerobically at 37 for 48-72 hours and aspectically streak the plates 19,20.
2. Identification of bacteria by culture characteristics ,microscopic examination and biochemical reaction 21.
3. Number of colony forming unit will be counted (CFU/ml)

ELIGIBILITY:
Inclusion Criteria:

* age group 4 -8 years.
* good health.
* No recent history of antibiotic coverage for at least two weeks
* necrotic teeth.
* restorable tooth structure.

Exclusion Criteria:

* more than 2/3 resorption of root.
* uncooperative patient.
* detection perforation on radiograph.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-05-12 (Actual)

PRIMARY OUTCOMES:
number of of colony forming units | 48 hours after culture
  number of of colony forming units less the better instrumentation technique and irritant

CONTACTS AND LOCATIONS:
Overall Officials: mansoura university, Study Chair — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Susila AV, Sai S, Sharma N, Balasubramaniam A, Veronica AK, Nivedhitha S. Can natural irrigants replace sodium hypochlorite? A systematic review. Clin Oral Investig. 2023 May;27(5):1831-1849. doi: 10.1007/s00784-023-04913-7. Epub 2023 Feb 18. PMID 36808559
- [Background] Sundaram D, Narayanan RK, Vadakkepurayil K. A Comparative Evaluation on Antimicrobial Effect of Honey, Neem Leaf Extract and Sodium Hypochlorite as Intracanal Irrigant: An Ex-Vivo Study. J Clin Diagn Res. 2016 Aug;10(8):ZC88-91. doi: 10.7860/JCDR/2016/19268.8311. Epub 2016 Aug 1. PMID 27656571
- [Background] Lakshmanan L, Jeevanandan G. Microbial Evaluation of Root Canals after Biomechanical Preparation with Manual K-files, Manual H-files, and Kedo-SG Blue Rotary Files: An In Vivo Study. Int J Clin Pediatr Dent. 2022 Nov-Dec;15(6):687-690. doi: 10.5005/jp-journals-10005-2457. PMID 36866149